CLINICAL TRIAL: NCT06292078
Title: Preventing School Exclusion and Opioid Misuse: Effectiveness of the Inclusive Skill-building Learning Approach (ISLA)
Acronym: ISLA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01DA059401-01 (NIH); 1R01DA059401-01 (NIH)
Record Dates: First submitted 2024-02-15; First posted 2024-03-04 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Middle Schools; School Exclusion; School Community; Teaching Practices; Opioid and Other Substance Misuse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Wave 1 Instructional Skill-Building Learning Approach (ISLA) (Experimental): Following a baseline year for data collection, school staff in 15 schools will be trained and supported in implementing ISLA schoolwide for two consecutive years.
  Interventions: Behavioral: Instructional Skill-Building Learning Approach (ISLA)
- Wave 1 Waitlist Control (No Intervention): These 15 schools will receive no intervention while wave 1 intervention schools undergo training and coaching on ISLA.
- Wave 2 Instructional Skill-Building Learning Approach (ISLA) (Experimental): Delayed one year after wave 1: Following a baseline year for data collection, school staff in 15 schools will be trained and supported in implementing ISLA schoolwide for two consecutive years.
  Interventions: Behavioral: Instructional Skill-Building Learning Approach (ISLA)
- Wave 2 Waitlist Control (No Intervention): These 15 schools will receive no intervention while wave 2 intervention schools undergo training and coaching on ISLA.

INTERVENTIONS:
Behavioral: Instructional Skill-Building Learning Approach (ISLA) — The Inclusive Skill-building Learning Approach (ISLA) is a school-wide, multi-component, instructional and restorative alternative to exclusionary discipline that begins with universal prevention grounded in positive, preventative classroom strategies for all students, and layers on additional supports for students in need.
  Arms: Wave 1 Instructional Skill-Building Learning Approach (ISLA); Wave 2 Instructional Skill-Building Learning Approach (ISLA)

SUMMARY:
This project will test the effectiveness of the Inclusive Skill-building Learning Approach (ISLA) in reducing the use of exclusionary discipline, improving teacher practice and student outcomes, and decreasing substance misuse using a randomized controlled trial in 60 middle schools across six states.

DETAILED DESCRIPTION:
Extensive research has documented the link between exclusionary discipline and numerous detrimental youth outcomes including lower academic achievement, a greater likelihood of being pushed out of school, and an increase in substance use and future criminal justice involvement. To engage in upstream prevention to reduce opioid and other substance misuse among youth there is a need to examine systems-wide, preventative interventions in schools to reduce educators biased and punitive interactions with students while implementing equitable supports. Thus, "Preventing School Exclusion and Opioid Misuse: Effectiveness of the Inclusive Skillbuilding Learning Approach (ISLA)" is being submitted to the National Institutes of Health, through the HEAL Initiative (RFA-DA-23-051). The proposed project aims to evaluate the effectiveness of ISLA, an instructional and restorative alternative to exclusionary discipline, on improving the social determinants of health (SDOH) of education access and quality, and social and community context to prevent school exclusion and opioid and other substance misuse. The investigators will conduct an effectiveness-implementation Hybrid Type 1 clustered randomized controlled trial in 60 middle schools across six states. All students and educators randomized to treatment will receive ISLA, and the investigators will evaluate impacts of ISLA on student outcomes from the end of 6th to the end of 8th grade. In addition, the investigators will incorporate methods to understand intervention processes across multiple levels of the school context. Our first aim is to examine the effectiveness of the ISLA. The investigators will test the direct effects of ISLA on the SDOH of education access and quality, specifically: (a) exclusionary discipline practices (office discipline referrals, in- and out-of-school suspensions, expulsions); (b) student engagement; and (c) inclusive teaching practices. The investigators will also test the direct effects of ISLA on the SDOH of social and community context, specifically: (a) student-teacher relationships; and (b) school climate. Additionally, the investigators will test the direct effects of ISLA on opioid and other substance misuse and associated risk factors. Our second aim is to examine the mediators and moderators of ISLA intervention effects which serve as key mechanisms for change in opioid and other substance misuse and associated risk factors. The investigators will examine the putative mediating effects of ISLA social determinant mechanisms on opioid and other substance misuse and associated risk factors. The investigators will also examine the potential moderating effect between student race/ethnicity and the ISLA intervention on reductions in exclusionary disciplinary practices. Finally, our third aim is to evaluate the implementation outcomes of the ISLA intervention, including: (a) feasibility, usability, acceptability, and fidelity; (b) sustainment; and (c) cost analysis. This project will fill a persistent gap in the field of substance use, by evaluating whether upstream school-based preventative interventions that target and improve SDOH can have meaningful impacts on preventing opioid and other substance misuse and associated risk factors.

ELIGIBILITY:
Teachers: The educator sample will include all educators within each of the schools. All educators that have regular contact with students (e.g., administrators, teachers, instructional assistants, school counselors) will participate in the school-wide ISLA intervention activities. All educators at both treatment and control schools, if they consent, will provide data through an annual survey administered at three time points: in the spring prior to the first year of ISLA implementation (baseline), in the spring of the first year of ISLA implementation (post-intervention), and in the spring of the second year of ISLA implementation (follow-up).

* Inclusion criteria:

  * Staff member in either a control or intervention condition school
* Exclusion criteria:

  * None

Cohort Students: The student cohort sample will include all students in Grade 7 during the first year of ISLA implementation, who will be followed into Grade 8 during the second year of ISLA implementation (such that data can be collected from the end of Grade 6 to the end of Grade 8). With an average middle school size of 660 students per school, we project the cohort size to be 220 students per school, for a total of 11,880 to 13,200 students.

Sub-cohort Students: A random sample of 50 assenting 6th grade students (at the time of baseline data collection) per cohort per school will be selected to provide additional data, for a total of 2,700 to 3,000 students (consent will be gathered from parents/guardians). With the help of each school administrator, the research team will conduct the randomization process using each school's enrollment. School administrators will invite all 6th grade students to participate via recruitment emails to their parents/guardians. A random selection of students will be made from those parents who are consented.

* Inclusion Criteria:

  * 6th grade students in either intervention or control schools during first data collection period for each wave
* Exclusion Criteria:

  * students who cannot complete the online survey independently (e.g., require assistance beyond text-to-speech files to comprehend the items and available responses) specifically:
  * students who cannot comprehend written or spoken English or written or spoken Spanish, or
  * students who are eligible for alternate assessment for statewide achievement testing.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5076 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Frequency and Duration of Use of Office Discipline Referrals, In-School Suspension, and Out-of-School Suspension | baseline, 1 year, 2 years
  We will collect data on the use of office discipline referrals (ODRs), in-school (ISS), and out-of-school suspensions (OSS). As part of the National TA Center on PBIS, all schools that will be recruited for this project use the School-Wide Information Systems (SWIS; May et al., 2013), a web-based behavior tracking platform, to enter and review behavior incidents and actions taken by school personnel including office discipline referrals (ODRs), in-school (ISS), and out-of-school suspensions (OSS).
Engagement vs. Disaffection with Learning Student-report | baseline, 1 year, 2 years
  The Engagement vs. Disaffection with Learning Student-report assesses engagement as a key component of motivated action leading to student learning and achievement. The assessment measures engagement versus disaffection in the classroom ranging from enthusiastic, effortful, emotionally positive interactions with learning activities to apathetic withdrawal and frustrated alienation, with both positive manifestations of behavioral and emotional participation in classroom and withdrawal of behavioral and emotional participation and alienation from learning. All items have five response options: (1) Not at all True; (2) A little True; (3) Mostly True; (4) Very True; (5) Prefer not to answer.
Inclusive Teaching Practices | baseline, 1 year, 2 years
  The WOW+ (Welcome at the door, Own your environment, Wrap up with intention +) Self-Report measures inclusive teaching practices, both general and specific teaching strategies that are part of the ISLA intervention. All school personnel in all treatment schools will receive training on the ISLA strategy for universal relationship building, known as the WOW strategy, which consists of three concrete skills rooted in behavioral science that educators can apply every day to create positive classroom environments: welcome students, own your classroom environment, and wrap up class with the intention. The WOW+ Self-Report is an adaption of the WOW Classroom Observation Tool which is a five-item measure with individual item scores ranging from 0 to 2, where each item is an operationally defined behavior based on the elements of the WOW strategy training.
School Climate Survey- Student | baseline, 1 year, 2 years
  The School Climate Survey: Secondary (SCS-S) is a 36-item, computerized school climate rating scale (Center on PBIS, 2022). The purpose of the SCS-S is to obtain middle and high school student perception ratings of school climate. Respondents use a 4-point Likert scale: 1=Strongly Disagree, 2 = Disagree, 3 = Agree, and 4 = Strongly Agree. To compute the overall school climate score, item responses are summed and then divided by the total number of items. Higher overall scores reflect a positive sense of the school environment with respect to (a) interpersonal relations among and between peers and adults, (b) learning environment, and (c) feelings of belonging and acceptance.
School Climate- Teacher | baseline, 1 year, 2 years
  The School Climate Survey: School Personnel (Center on PBIS, 2022) includes 29 items and 5 subscales, including staff connectedness, structure for learning, school safety, physical environment, peer and adult relations, and parent involvement. School personnel rate items as Strongly Agree, Somewhat Disagree, Somewhat Agree or Strongly Agree. The personnel survey also demonstrates adequate psychometric properties with an internal consistency of .94 for the overall school climate scale.
Student-Teacher Relationships | baseline, 1 year, 2 years
  The Adult Social Support subscale from the School Climate Survey: Student (SCS-S; Center on PBIS, 2022) will be used to measure student-teacher relationships in schools. The Adult Social Support subscale contains four items and has strong internal consistency (α = .91). A high mean score on the Adult Social Support subscale represents a positive feeling of adult support and encouragement, whereas a low score suggests poor interpersonal relationships among students and adults within the school. From this subscale, we expect to understand data about student engagement, school climate, opioid and other substance misuse, internalizing and externalizing behaviors.
Opioid and Other Substance Misuse | baseline, 1 year, 2 years
  Thirteen opioid and other substance misuse questions and response criteria are derived from the Monitoring the Future survey conducted annually with adolescent youth throughout the United States and the National Institute on Drug Abuse-modified Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) measure. The survey is funded by NIDA as an on-going surveillance effort to understand and report substance use trends among youth. Respondents use an ordinal response scale with seven options (0 Occasions; 1-2; 3-5; 6-9; 10-19; 20-39; 40 or more) to describe substance use during the last 12 months.
Student Internalizing Behaviors | baseline, 1 year, 2 years
  The Strengths and Difficulties Questionnaire (SDQ; Goodman 1997) is a brief (25 items) behavioral screening questionnaire about psychosocial problems for youth, and includes competencies or strengths in addition to assessing problems. The SDQ is equally divided across five scales measuring emotional symptoms, conduct problems, hyperactivity-inattention, peer problems, and prosocial behavior. Participants rate items as Not True, Somewhat True, or Certainly True. The SDQ has adequate psychometric properties with internal consistency of .68 and test-retest reliability of .62.
Student Externalizing Behaviors | baseline, 1 year, 2 years
  Nine items from the Youth Self-Report (YSR; Achenbach, 1991) will be used to measure student externalizing behaviors. The YSR asks students now or within the past 6 months, how often they had the following problems: Hangs around bad kids; Swears; Uses alcohol or drugs; Truant; Runs away; Lies or cheats; Prefers older kids; Doesn't feel guilty. Each item has three categories: 0 = not true or not at all, 1 = sometimes or somewhat true, or 2 = very true or often. The internal consistency of these items was α = .68 (Song et al., 1994).
ISLA Acceptability | 1 year and 2 years for intervention condition schools
  The Primary Intervention Rating Scale (PIRS) will be used as a measure of the feasibility, usability, and acceptability of the ISLA intervention by gathering educator perceptions of the social validity of intervention goals and procedures (Lane et al., 2002). The PIRS is a 17-item survey completed on a Likert scale with allowable responses of Strongly Disagree, Disagree, Slightly Disagree, Slightly Agree, Agree, and Strongly Agree. The PIRS has adequate psychometric properties, with internal consistency of .97, and the correlation between schools' PIRS scores and treatment integrity scores was r = .71 (Lane et al., 2009). To the PIRS we have added two items relating to sustainment, and four open-ended items that have been applied in previous research (Furjanic et al., 2021).
ISLA Implementation Fidelity | baseline, 1 year, 2 years
  The fidelity if ISLA implementation will be measured using student-level ISLA fidelity tracking sheets (maintained by the ISLA support staff member in each school), and the school-wide ISLA Implementation Checklist (completed by the school team). The ISLA fidelity tracking sheet is used to record information about each student that accesses the ISLA support room, and the ISLA support staff completes Yes/No questions about ISLA delivery for each student.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Soquel Union Elementary School District, Capitola, California
  - Riverbend School District, Yuba City, California
  - Salem-Keizer School District, Salem, Oregon